CLINICAL TRIAL: NCT06263842
Title: Peri-implant Clinical and Radiographic Alterations Following Immediately Placed, Immediately Loaded Dental Implants Using Socket Shield Approach With Autogenous Whole Tooth Graft Versus Xenograft: Randomized Clinical Tial
Brief Title: Elamrousy Novel Approach of Socket Shield Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-132
Record Dates: First submitted 2024-02-07; First posted 2024-02-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Implant Complication
MeSH Terms: interventions — Immediate Dental Implant Loading; Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: The present study included 63 participants, aged 20 to 45, with teeth that needed to be extracted. After Kafrelsheikh University research ethics committee approval, patients were randomized into 3 groups: group I patients underwent immediate implantation using SSA protocol without grafting, while group II was grafted by xenograft, but group II was grafted with AWTG was created using the decoronated crown and the extracted palatal portion of the tooth; and then placed in the peri-implant gap defect. Clinically, pink aesthetic score (PES), midfacial mucosal alterations (MFMA), stability quotient of dental implants (SQDI) were observed at baseline, six and twelve months after implantation. Moreover, baseline, 6- and 12-months alterations of radiographic horizontal buccolingual ridge width (HBLRW), facial marginal bone level (FMBL), peri-implant Density of bone (PIDB) and peri-implant vertical bone defect depth (PIVBDD) changes were assessed using cone beam computed tomography (CBCT).
Who Masked: Participant, Outcomes Assessor
Masking Description: neither participant nor the outcome assessor know the group distribution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Implant Placement Using Socket Shield Technique alone (Experimental): after insertion of immediate implant Using Socket Shield Technique, the bone defect between the socket shield and the implant fixture will be left ungrafted
  Interventions: Procedure: conventional socket shield
- Immediate Implant Placement Using Socket Shield Technique with xenograft (Experimental): the shield/fixture jumping gap will be grafted with xenograft
  Interventions: Procedure: combined socket shild with xenograft
- Modified Elamrousy Approach for Immediate Implant Placement Using Socket Shield Technique (Experimental): Immediate Implant Placement Using Socket Shield Technique with autogenous whole tooth graft after immediate implantation using Socket Shield Technique, the palatal root portion and the decoronated crown will be converted to autogenous whole tooth graft and used for grafting the defect between the socket shield and the implant fixture
  Interventions: Procedure: modified Elamrousy approach for socket shield technique

INTERVENTIONS:
Procedure: modified Elamrousy approach for socket shield technique — the jumping gap will be filled with AWTG
  Arms: Modified Elamrousy Approach for Immediate Implant Placement Using Socket Shield Technique
Procedure: conventional socket shield — the jumping gap will be left ungrafted
  Arms: Immediate Implant Placement Using Socket Shield Technique alone
Procedure: combined socket shild with xenograft — the jumping gap will be filled with xenograft
  Arms: Immediate Implant Placement Using Socket Shield Technique with xenograft

SUMMARY:
The current trial aim was to evaluate clinically and radiographically the changes around dental implants inserted immediately in maxillary anterior esthetic zone using a novel combination of autogenous whole tooth graft (AWTG) with socket shield approach (SSA) and compared this approach to socket shield technique with xenograft.

The present study included 63 patients, aged 20 to 45, with teeth that needed to be extracted. After Kafrelsheikh University research ethics committee approval, patients were randomized into 3 groups: group I patients underwent immediate implantation using socket shield protocol, while group II patients underwent the same procedure, but the shield/fixture jumping gap was grafted by xenograft. finally group III was grafted by AWTG that was created using the decoronated crown and the extracted palatal portion of the tooth; and then placed in the peri-implant gap defect.

DETAILED DESCRIPTION:
It has been demonstrated that utilizing dental implants to replace lost teeth is a predictable clinical choice. Promising outcomes of immediate implant insertion in conjunction with immediate loading/provisionalization (Type 1A implant protocol according to Gallucci et al has been reported to provide major benefits in terms of better esthetic and psychosocial impacts, shorter treatment duration, minimal surgical interventions and preservation of peri-implant bone and soft tissue.

However, because of technically sensitive and sophisticated surgery required for Type 1A protocol, high risk of early implant failure was noticed particularly in conditions that might complicate that protocol as deficient facial bone plate, soft tissues deficiencies and thin gingival phenotype. Furthermore, those conditions also were found to be responsible for midfacial mucosal recession (MFMR), papillary recession and resorption of facial plate that deteriorates the clinical, radiological, and esthetic outcomes of Type 1A protocol. Consequently, alternate approaches would be suggested to improve the clinical and esthetic concerns associated with immediate implantation and loading such as buccal gap grafting, guided bone regeneration and socket shield approach.

In order to maintain the facial bone plate for prompt Type 1A protocol in esthetic zone, the SSA has been developed by Hürzeler et al. in 2010 as a potential therapeutic approach through maintaining the facial portion of the root and thus preserving the periodontal ligament and its vascularity that nourishes the tooth's bundle bone. The FSS functions as a natural barrier that prevents buccal bone resorption and enhances tissue contouring, both of which contribute to the achievement of predictable esthetic outcomes. Additionally, the FSS serves as a guide to ensure the implant is positioned correctly. SSA in conjunction with immediate loading reduces the frequency of clinical sessions and reduces the necessity for both soft and hard tissue grafts.

It has been recommended to palatally insert the implants in extraction sockets with at least 2 mm jumping gap between the fixture and the FSS. Significantly, this gap denotes the future buccal bone that will directly contribute to the buccal contour and impact the soft tissue levels. For jumping gaps smaller than 2 mm, bone heals spontaneously, while gaps bigger than 2 mm are advised to be augmented.

AWTG is obviously very advantageous as it exhibits superior osteoconductive and osteoinductive capacity with high biocompatibility and comparable physico-chemical characteristics to autogenous bones. AWTG was successfully employed for augmenting of peri-implant bone defects, with excellent clinical and radiographic outcomes. Similarly, both AWTG and autogenous demineralized dentin graft were equally effective at reducing dimensional losses in alveolar ridge preservation. The production of demineralized dentin is time-consuming, cost-intensive and complicated, which restricts its widespread use in clinics.

In the light of this, the current study was conducted to assess and compare the effectiveness of AWTG versus xenograft for augmenting the FSS/fixture jumping gap around immediately placed implants using SSA with immediate temporization in the maxillary esthetic zone.

To the best of our knowledge, this study is the first to use AWTG for filling the peri-implant jumping gap following SSA and highlight its impact on peri-implant soft and hard tissue parameters compared to xenograft.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 18years
* presence of non-restorable maxillary anterior tooth
* had sufficient bone volume and
* The primary stability at insertion not less than 35 N

Exclusion Criteria:

* history of systemic condition
* history of using bisphosphonates or other drugs that might impact bone turnover
* a history of smoking during the previous five years,
* a history of any acute infections at the surgical site,
* teeth having root resorptions
* massive periodontal destruction

  , the presence of any systemic diseases;
* intake of drugs that may alter bone metabolism
* presence of acute infection
* infra-bony horizontal tooth fracture
* facial vertical root fracture;
* root resorption; mobile teeth
* malaligned teeth,
* active periodontitis at the implantation site.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Stability Quotient of dental implant (SQDI) | 12-month.
  Osstell TM was used to record the primary stability.ISQ, or Implant Stability Quotient, is a scale from 1 to 100 and is a measure of the stability of an implant. The ISQ scale has a non-linear correlation to micro mobility. With more than 1400 scientific references, investigators now know that high stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
pink esthetic score (PES) | 12-month.
  The pink esthetic score (PES) evaluates the esthetic outcome of soft tissue around implant-supported single crowns in the anterior zone by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency.Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES was 14
Midfacial Mucosal Alterations | 12-month.
  digital intraoral scans were recorded. To quantify the vertical changes in the soft tissues around implants buccally, the collected scans were digitally superimposed via matching Gom inspect software

SECONDARY OUTCOMES:
facial marginal bone level (FMBL) | 12-month.
  Utilizing CBCT sagittal sections, the BMBL was evaluated by computerized analysis. Navigation was done on the multiplanar display until the implant's precise same-view location was established on the reformatted cross-sectional section and panoramic view.

CONTACTS AND LOCATIONS:
Overall Officials: Walid AH Elamrousy, PhD, Principal Investigator — Faculty of Oral and Dental Medicine, Kafrelsheikh University
Locations (1):
- Walid Elamrousy, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers